CLINICAL TRIAL: NCT04210050
Title: Implementation of a Precision Sleep Ventilation (PSV) Chronic Respiratory Failure Management Program for Patients With Advanced Hypercapnic COPD
Brief Title: Sleep Ventilation for Patients With Advanced Hypercapnic COPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was not initiated due to COVID19 pandemic
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Breas Medical S.A.R.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P000778
Record Dates: First submitted 2019-12-17; First posted 2019-12-24 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Blood Gas Analysis

STUDY DESIGN:
Intervention Model Description: The model is a prospective, randomized, comparative effectiveness clinical trial to evaluate the role of non-invasive nocturnal ventilation in addition to usual care, compared to usual care alone in the management of adult COPD patients with chronic hypercapnic respiratory failure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual care (Other): Usual care follows the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines.
  Interventions: Diagnostic Test: Arterial blood gas (ABG) and serum bicarbonate level; Diagnostic Test: Overnight home oximetry and transcutaneous CO2 monitoring
- Usual care plus NIPPV group only (Active Comparator): Usual care for COPD based on Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines plus use of nocturnal ventilator device using the Breas VIVO 50 home ventilator, Breas Medical (or any newer models as available).
  Interventions: Device: Home noninvasive nocturnal ventilation with Breas VIVO 50 home ventilator or newer model as available, Breas Medical.; Diagnostic Test: Arterial blood gas (ABG) and serum bicarbonate level; Diagnostic Test: Overnight home oximetry and transcutaneous CO2 monitoring

INTERVENTIONS:
Device: Home noninvasive nocturnal ventilation with Breas VIVO 50 home ventilator or newer model as available, Breas Medical. — In the usual care plus NIPPV group, those able to undergo attended PSG will be titrated with volume targeted pressure support mode, aiming to lower the baseline TcCO2 by 10 mmHg. In some cases, the CO2 cannot be lowered by that amount on a single titration, but rather will decrease over time.
  For those unable to undergo lab titration (too frail, no transportation, decline/refuse), NIPPV will be initiated with empiric settings based on nighttime home CO2 tracking and daytime ABG monitoring.
  Arms: Usual care plus NIPPV group only
Diagnostic Test: Arterial blood gas (ABG) and serum bicarbonate level — Will be obtained at baseline (before randomization), then at 3, 6 and 12 months into the study
Diagnostic Test: Overnight home oximetry and transcutaneous CO2 monitoring — will be conducted at 1 and 6 months into the study (for subjects in the NIPPV plus usual care group, testing will be done while using the ventilator.

SUMMARY:
Despite growing evidence showing benefit (in both clinical and cost standpoints), only a small percentage of COPD patients with chronic hypercapnic respiratory failure are managed with nocturnal ventilatory support. There is uncertainty of the value of aggressive nocturnal ventilation, especially polysomnographic estimation of therapy and home transcutaneous CO2 tracking.

The driving goal behind this project is to develop and implement a streamlined and comprehensive program for nocturnal ventilator management of patients with advanced, hypercapnic COPD.

DETAILED DESCRIPTION:
The purpose of this protocol is to perform a prospective, randomized, comparative effectiveness clinical trial to evaluate the role of non-invasive nocturnal ventilation in addition to usual care, compared to usual care alone in the management of adult COPD patients with chronic hypercapnic respiratory failure. The study will focus on the primary end-points of time to hospital re-admission for acute exacerbation of COPD and/or an episode of acute on chronic hypercapnic respiratory failure, in addition to other clinically relevant outcomes including patient health-related quality of life, sleep quality indices, and gas exchange parameters. Approximately 300 BIDMC adult patients will be recruited and each patient monitored over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure.
2. Male or female aged ≥ 18 years with advanced hypercapnic COPD

   1. FEV1 ≤ 50% predicted and
   2. Prolonged hypercapnia during the daytime, at rest, without O2 or ventilatory support, PaCO2 > 52 mmHg on ABG (performed off of NIPPV), compensated with pH > 7.30
3. Willingness to use NIPPV treatment
4. English speaking

Women and minorities will be recruited in numbers reflecting representation in the Boston Metropolitan community which is approximately 84% Caucasian, 9% African American, 5% Hispanic American, and 2% Asian American, as the knowledge gained can apply to individuals of all ethnic background and gender.

We do not wish to limit our sample to a highly selected group of patients, to allow for more generalizable results.

Exclusion Criteria:

Subjects will be excluded from participation in the study for a history of:

* Significant sleep disordered breathing (AHI 4% ≥ 15 events/hour) or high clinical suspicion (BMI ≥ 35)
* Neuromuscular disease or other causes of hypoventilation
* Abnormalities of the thorax or lungs other than COPD
* Already treated with home NIPPV
* Unable to wean from ventilator during admission
* Unable to wean from NIPPV, pH < 7.30
* Recent tracheotomy decannulation
* History of severe depression or bipolar disorder requiring prior hospitalization or suicide attempts or ideation
* Cognitive impairment (such as advanced dementia) that would limit ability to provide consent or to use NIPPV
* Active recreational drug use
* Unstable housing that would limit ability to use NIPPV
* Severe heart failure (New York Heart Association stage IV)
* Active/unstable CAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time to readmission or death | within 12 months
  time to re-admission for acute exacerbation of COPD and/or acute on chronic hypercapnic respiratory failure or death

SECONDARY OUTCOMES:
Patient health related quality of life (HRQOL) | 12 months
  The RAND SF-36, a 36-question multiple choice QOL form will be used to assess general health perception. The questions target eight health domains or scales: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal/emotional problems, emotional well-being, social functioning, energy/fatigue, general health perceptions, and one's perceived change in health.
  There is a 2-step process used in scoring, such that the score for each of the scales represent the average for all item in the scale that were answered. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Next, items in the same scale are averaged together to create 8 scale scores. The lower the score the more disability and the higher the score the less disability.
  Scores will be assessed at baseline, 3 and 12 months for usual care and usual care plus ventilation support for all subjects.
Dyspnea scale | 12 months
  change in results of the Medical Research Council dyspnea scale, a categorical scale from 1-5, higher score =more limitation on daily activity due to breathlessness. Scores will be assessed at baseline, 3 and 12 months for usual care and usual care plus ventilation subjects.
Gas exchange | 12 months
  Change in CO2 from ABG and serum bicarbonate
General health status | 12 months
  St. George's Respiratory questionnaire, a 50 item questionnaire that measures health status in patients with COPD will be completed at baseline, and after 3 and 12 months in all subjects. For this questionnaire, a score of 0 = best QOL, and a score of 100 = worst QOL. The questions focus on three areas - symptoms, activity, and impact (psycho-social).

OTHER OUTCOMES:
Ambulatory BP profiles | 3 months compared to baseline
  In a subset of subjects (from usual care and usual care plus ventilation groups), 24-hour ambulatory BP monitoring will be conducted (at baseline and after 3 months) to assess for change in 24-hour and nocturnal systolic, diastolic and mean BPs.
Inflammatory biomarkers | 3 and 12 months compared to baseline
  High sensitivity C-reactive protein [hs-CRP], units mg/ml, can be measured from peripheral blood. Elevated levels reflect increased systemic inflammation. Studies have shown that individuals with elevated levels (above 2 mg/ml) are at increased risk of cardiovascular disease. During this trial, HR-CRP will be obtained at baseline and after 3 and 12 months in subjects to assess whether there is a favorable change in subjects treated with nocturnal ventilation + usual care, as compared to usual care.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Subject information and biological samples will be used and shared with the researchers involved in this study to conduct the research.